CLINICAL TRIAL: NCT02226237
Title: URINARY INCONTINENCE AND ERECTIL DYSFUNCTION AFTER RADICAL PROSTATECTOMY: A Randomized Controlled Trial Comparing Pelvic Muscle Exercises With or Without Electrical Stimulation
Brief Title: Effectiveness of Physiotherapy to Treat the Urinary Incontinence and Erectile Dysfunction Post Retropubic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Wesley Justino Magnabosco, MD, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSTXPTR2010
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Incontinence; Erectile Dysfunction
Keywords: urinary incontinence; erectile dysfunction; Retropubic Prostatectomy; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): in which patients received no specific treatment, only the usual general guidelines
- group of pelvic floor exercises (Experimental): in which patients were instructed to perform home exercises daily
  Interventions: Procedure: group of pelvic floor exercises
- anal electrostimulation group (Experimental): in which patients, and are instructed to perform the exercises mentioned in the group of pelvic floor exercises, also underwent anal electrostimulation
  Interventions: Procedure: group of pelvic floor exercises; Procedure: anal electrostimulation group

INTERVENTIONS:
Procedure: group of pelvic floor exercises — contraction of the pelvic floor muscles sustained for 5 seconds, hip adductors using pillow and elevation of the hip, 30 repetitions of each exercise
  Arms: anal electrostimulation group; group of pelvic floor exercises
Procedure: anal electrostimulation group — The anal electrical stimulation protocol was performed by a physical therapist for seven weeks, twice per week, using the apparatus Dualpex 961 Uro® Quark, with frequency of 35 Hz, and the intensity determined according to the tolerance of the patient, lasting 20 minutes.
  Arms: anal electrostimulation group

SUMMARY:
The prostate cancer is the most common parenchymal neoplasia in men over 45 years old. Radical prostatectomy is curative treatment is most used today. Urinary incontinence and erectile dysfunction are the main complications of radical prostatectomy. Physical therapy has been used as a form of conservative treatment of these complications. However, the role of physiotherapy in the treatment of these complications is not well defined in the literature. We will do a randomized controlled study with patients undergoing radical prostatectomy. After removal of the Foley catheter, patients will be randomized into 3 groups: control group, group of pelvic floor exercises and anal electrostimulation group. These patients will be evaluated preoperatively in an attempt to meet prognostic factors for urinary incontinence and erectile dysfunction. They will be followed by 2 years after surgery, to assess whether the therapy will alter the course of urinary continence and erectile function in these patients.

DETAILED DESCRIPTION:
Randomization was performed by a team of external statistics to the research team, using the method of randomization in blocks of three, who were randomly selected. The group to which the patient was allocated to researchers only be informed at the time of randomization, if patients satisfied the criteria for inclusion and exclusion.

Will be evaluated preoperatively: urodynamic studies and clinical evaluation. The following clinical data were evaluated: Body Mass Index (BMI), comorbidities, disease staging and sociodemographic information.

The following parameters will be evaluated in the pre-operative and after one, three, six and twelve months after surgery: evaluating the strength of the pelvic floor through perineometry, the 1 hour pad test, electromyographic evaluation of pelvic floor, and the application of instruments validated for the Portuguese language. The follow instruments will be applied: International Index of Erectile Function - 5 questions (IIEF-5), International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), International Prostate Symptom Score (IPSS).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* diagnosed with localized or locally advanced prostate cancer
* that are undergoing radical prostatectomy as treatment of the condition
* they are coming from Barretos or a nearby region or has logistics facilities to come to the Barretos Cancer Hospital to perform the followup

Exclusion Criteria:

* those with mental or physical problems that make it impossible to collect data or that may influence the recovery of continence postoperatively
* patients with metastatic prostate cancer
* patients not undergoing retropubic prostatectomy as treatment for prostate cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
recovery of urinary continence | one year
recovery of erectile function | two years

SECONDARY OUTCOMES:
evaluate prognosis for recovery of urinary continence | one year
  assess the presence of prognostic factors for the recovery of urinary continence after radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Wesley J Magnabosco, MD, Principal Investigator — Barretos Cancer Hospital; João L Amaro, PhDh, Study Director — UPECLIN HC FM Botucatu Unesp; Carla LC Andrade, Principal Investigator — Barretos Cancer Hospital; Fernanda Jabur, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo State, Brazil

REFERENCES:
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660